CLINICAL TRIAL: NCT02147366
Title: Role of Music in Non Pharmacological Management of Hypertension
Brief Title: Indian Instrumental Music in Hypertension
Acronym: MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MS Ramaiah Medical College & Hospitals (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, KIRTHANA KUNIKULLAYA U, Dr. Kirthana Kunikullaya U, Assistant Professor, MS Ramaiah Medical College & Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-13440
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Hypertension,ambulatory pressure,autonomic function,music
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral (Lifestyle) (Experimental): Only standard lifestyle modifications The prehypertensives and stage I hypertensives will be randomized to receive each of the two three experimental conditions: music along with standard lifestyle modifications or only standard lifestyle modifications in random order over the course of three months.
  Interventions: Behavioral: Lifestyle
- Behavioral (Music & lifestyle changes) (Experimental): Experimental: Music along with standard lifestyle modifications The prehypertensives and stage I hypertensives will be randomized to receive each of the two three experimental conditions: music along with standard lifestyle modifications or only standard lifestyle modifications in random order over the course of three months.
  Interventions: Behavioral: Music & lifestyle changes

INTERVENTIONS:
Behavioral: Music & lifestyle changes — Music intervention involved listening to raga bhimpalas played on bansuri/flute (an Indian instrument) for 15 minutes daily for 3 months.
  Arms: Behavioral (Music & lifestyle changes)
Behavioral: Lifestyle — Lifestyle intervention was based on Joint national committee VII guidelines for hypertension
  Arms: Behavioral (Lifestyle)

SUMMARY:
* Hypertension is one of the leading risk factors influencing morbidity and mortality. There is need for non-pharmacological management for the same. Music is known to reduce anxiety and holds promise for non-pharmacological management of hypertension owing to low cost, ease of administration and safety. The efficacy of music to reduce blood pressure (BP) has not been established. Besides inconsistent findings, earlier studies using music are frequently inconclusive from small sample size. The studies have not examined the biomarkers of hypertension.
* The purpose of this study was to evaluate the effect of Indian Instrumental music on pre-hypertensives and stage 1 hypertensives subjects. Non-pharmacological intervention improves the quality of life of hypertensives and music may serve as an adjunct therapy along with standard management of hypertensives.

DETAILED DESCRIPTION:
Arterial hypertension is an important risk factor for diseases like myocardial infarction and stroke leading to increased morbidity and mortality. Lifestyle modifications are often recommended as a part of treatment for mild hypertension, but the efficacy of the adjunct therapy is unclear. Weight loss and salt restriction are the most effective modalities, but each requires a major change in dietary habits, which is difficult for patient compliance.

A number of therapeutic modalities that aim to reduce stress and encourage relaxation have been evaluated for the treatment of hypertension. Various methods like autogenic training, cognitive therapy, behavioral therapy, Meditation, Guided imagery, biofeedback, progressive muscle relaxation, breathing exercises, yoga have been previously studied to reduce hypertension.

Music has long been known to reduce anxiety, minimize the need for sedatives, and make patients feel more at ease. Music therapy is different from music medicine. Music therapists individualize their interventions according to patient's needs. Patients actively get engaged in music making. However, in music medicine, subject listens to pre-recorded music with perceived benefit.

A number of research studies have been conducted to determine the effects of music on a variety of clinical conditions. Effect of music on stress reduction has been documented in physiological (e.g. heart rate, blood pressure), neurological (e.g. EEG readings) and psychological domains. In addition, the effect of music intervention has been documented in a range of medical, surgical, oncology, and pediatric patients.

In one of the studies on hypertensive individuals, there was a significant decrease in both systolic (15.9 mm Hg reduction) and diastolic BP (9 mm Hg) after weekly music therapy sessions for duration of 12 weeks. The control group did not show significant changes (Márquez-Celedonio, 2009). Among hypertensives, there was a significant reduction in BP after using a device which guides the user towards slow and regular breathing using musical sound patterns. The device was used for 10 minutes daily at home for 8 weeks. The control group in this study were given a walkman with which patients listened to quiet music. Treatment with the device reduced systolic BP, diastolic BP and Mean arterial pressure (MAP) by 15.2,10.0 and 11.7 mm Hg respectively, as compared to 11.3, 5.6 and 7.5 mm Hg with the Walkman (Schein, 2001). Another study evaluated the short and long-term effects of audio relaxation programs for BP reduction in older adults. The subjects listened to a 12-minute audio relaxation program. The reduction in systolic and diastolic BP was statistically and clinically significant (Tang, 1996).

There are very few studies that have examined the effect of music on hormone levels that are of particular relevance to heart disease, including adrenaline and noradrenaline concentrations levels and other stress hormones that can be deleterious to cardiac functioning. Further, to the best of our knowledge, there are no studies done among prehypertensives using music as the intervention.

Thus we propose to study whether blood pressure among prehypertensives and stage 1 hypertensives can decrease after music intervention. In order to know the mechanism underlying this reduction, we propose to study the biomarkers (indicating the function of vascular endothelium, stress hormones, oxidative stress) responsible in the causation of hypertension and autonomic function. A better understanding of alterations in these biomarkers will help us to explain the mechanism of action and validate music intervention as a tool in non-pharmacological management of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* age group of 30 to 60 years. Prehypertensives and stage I hypertensives were identified as per Joint National Committee (JNC) VII classification

Exclusion Criteria:

* Pregnant women, subjects with body mass index (BMI) ≥35 kg/m2, stage 2 Hypertension (HTN), renal impairment, uncontrolled diabetes, raised intracranial tension, stroke, epilepsy, hearing problems, psychiatric disorder, other cardiovascular and respiratory disorders, or any other illness which is known to affect the BP status of the individual were excluded from the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
24 hour Blood Pressure | 3 months
  Blood Pressure in mm of Hg - Overall, awake and asleep

SECONDARY OUTCOMES:
Biomarkers of hypertension | 3 months
  Plasma catecholamines, renin, endothelin and superoxide dismutase
Autonomic function | 3 months
  Heart rate variability parameters (Time domain and frequency domain)

CONTACTS AND LOCATIONS:
Overall Officials: KIRTHANA U KUNIKULLAYA, MD, DNB, Principal Investigator — M S Ramaiah Medical college and hospitals
Locations (1):
- M S Ramaiah Medical college and hospitals, Bangalore, Karnataka, India